CLINICAL TRIAL: NCT06090123
Title: A Phase 1,Parallel Assignment,Fixed-Sequence Study to Assess the Effect of Itraconazole, Rifampicin on the Pharmacokinetics of TPN171H in Healthy Subjects
Brief Title: Drug-Drug Interaction (DDI) Study for TPN171H
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPN171H-05
Record Dates: First submitted 2023-06-21; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPN171H and Itraconazole (Experimental): Single dose of 10mg TPN171H on Day 1, 200mg Itraconazole(QD) on Days 3-5, 10mg TPN171H and 200mg Itraconazole on Day 6.
  Interventions: Drug: TPN171H; Drug: Itraconazole
- TPN171H and Rifampicin (Experimental): Single dose of 20mg TPN171H on Day 1, 600mg Rifampicin(QD) on Days 3-9, 20mg TPN171H and 600mg Rifampicin on Day 10.
  Interventions: Drug: TPN171H; Drug: Rifampicin

INTERVENTIONS:
Drug: TPN171H — Sequence 1：Single dose of 10mg TPN171H on Day 1, 200mg Itraconazole(QD) on Days 3-5, 10mg TPN171H and 200mg Itraconazole on Day 6.
  Sequence 2：Single dose of 20mg TPN171H on Day 1, 600mg Rifampicin(QD) on Days 3-9, 20mg TPN171H and 600mg Rifampicin on Day 10.
Drug: Itraconazole — Sequence 1：Single dose of 10mg TPN171H on Day 1, 200mg Itraconazole(QD) on Days 3-5, 10mg TPN171H and 200mg Itraconazole on Day 6.
  Arms: TPN171H and Itraconazole
Drug: Rifampicin — Sequence 2：Single dose of 20mg TPN171H on Day 1, 600mg Rifampicin(QD) on Days 3-9, 20mg TPN171H and 600mg Rifampicin on Day 10.
  Arms: TPN171H and Rifampicin

SUMMARY:
The primary objective of this study was to assess the effect of rifampicin,a cytochrome P450 3A4 enzyme (CYP3A4) induction, on the pharmacokinetics (PK) of TPN171H in chinese healthy male subjects ,and assess the effect of itraconazole，cytochrome P450 3A4 enzyme (CYP3A4) induction on the PK of TPN171H in chinese healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 40 years;
2. Body Mass Index of 19 to 26 kg/m2; Body weight no less than 50 kg;
3. Physical examination, vital signs examination, ECG, laboratory examination results were normal or abnormal without clinical significance;
4. Take reliable contraceptive measures during the trial and within three months after taking the drug;
5. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the written informed consent, and can complete the whole trial process according to the test requirements.

Exclusion Criteria:

1. Allergies to test preparations, any of their ingredients, and related preparations; With allergies or allergic diseases;
2. Clear diseases of the central nervous system, cardiovascular system, digestive system (including those with severe fatty liver in B-ultrasound examination), respiratory system, urinary system, blood system, metabolic disorders, etc. and require medical intervention or other unsuitable clinical trials Those with tested diseases (such as history of mental illness, etc.); those with a history of orthostatic hypotension;
3. Blurred vision or a history of the following ocular diseases: nonvascular anterior ischemic optic neuropathy (NAION), abnormal color vision, hereditary retinal degeneration (such as retinitis pigmentosa), macular degeneration;
4. A history of postural hypotension;
5. Patients with blood loss ≥400 mL within 3 months before inclusion;
6. Taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health care products within 2 weeks before administration;
7. Participated in other drug clinical trials and received trial drugs within 3 months before administration;
8. Positive results of alcohol breath test, or current/previous alcoholics (drinking more than 21 standard units per week. 1 standard unit contains 14 g of alcohol, such as 360 mL of beer or 45 mL of 40% spirits or 150 mL wine);
9. Smoking more than 10 cigarettes per day ;
10. Positive for hepatitis B surface antigen (HBsAg), HCV antibody, syphilis antibody and HIV antibody;
11. Patients with clinically significant Chest x-ray (posterioranterior) abnormalities;
12. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Cmax of TPN171H | 48 hours after taking TPN171H
  Maximum Plasma Concentration (Cmax) of TPN171H
AUC of TPN171H | 48 hours after taking TPN171H
  Area under the plasma concentration versus time curve (AUC) of TPN171H

SECONDARY OUTCOMES:
Adverse events | Up to Day 13 from taking TPN171H for part one(Itraconazole), up to Day 17 from taking TPN171H for part two(Rifampicin)
  Number of Participants With treatment-related Adverse Events and Serious Adverse Events
The pharmacokinetic parameters (TPN171H) :Tmax | 48 hours after taking TPN171H
  The pharmacokinetic parameters (TPN171H) :Tmax
The pharmacokinetic parameters (TPN171H) :T1/2 | 48 hours after taking TPN171H
  The pharmacokinetic parameters (TPN171H) :T1/2
The pharmacokinetic parameters (TPN171H) :CL/F | 48 hours after taking TPN171H
  The pharmacokinetic parameters (TPN171H) :CL/F
The pharmacokinetic parameters (TPN171H) :Vz/F | 48 hours after taking TPN171H
  The pharmacokinetic parameters (TPN171H) :Vz/F

CONTACTS AND LOCATIONS:
Overall Officials: Gangyi Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No